CLINICAL TRIAL: NCT03609307
Title: Comparison of Treatment Response to Intravitreal Injection of Combined Propranolol and Bevacizumab Versus Bevacizumab Monotherapy in Patients With Wet Age Related Macular Degeneration :A Clinical Trial
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Clinical Professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 96301
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- injection Combined Intravitreal bevacizumab and propranolol (Active Comparator): patients receive two injections at each session Bavacizumab
  Interventions: Drug: Combined Intravitreal bevacizumab and propranolol
- injection Intravitreal bevacizumab (Active Comparator): patients receive only Bevacizumab
  Interventions: Drug: Intravitreal bevacizumab

INTERVENTIONS:
Drug: Combined Intravitreal bevacizumab and propranolol — these patients receive two injections at each session Bavacizumab and propranolol
  Arms: injection Combined Intravitreal bevacizumab and propranolol
Drug: Intravitreal bevacizumab — these patients receive only Bevacizumab
  Arms: injection Intravitreal bevacizumab

SUMMARY:
This study is designed to compare the effect of combined intravitreal Bevacizumab and Propranolol injection versus Bevacizumab monotherapy in patients with Age Related Macular Degeneration.

Methods:

In this study patients with Age Related Macular Degeneration who are naïve or had history of previous treatment are included. The eligible patients in randomized in two groups "Bevacizumab" and "Bavacizumab + propranolol" and in injected intravitreally for 3 times monthly. In "Bevacizumab+propranolol" group patients receive two injections at each session Bavacizumab and propranolol. In "Bevacizumab" group patients receive only Bevacizumab. The patients are followed for 6 months and central macular thickness and visual acuity is measured at baseline and monthly for 6 month. Baseline ancillary exams include Fluorescein Angiography and OCT-Angiography which is performed at the final exam as well. Patients needing any therapeutic intervention is addressed during the 6 month follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Wet AMD and Vision less than 20/40

Exclusion Criteria:

* History of cardiac ,renal, respiratory diseases (due to beta blocker toxicity),
* Associated with other Macular abnormalities such as Diabetic Retinopathy, Macular traction
* History of ocular inflammation
* Subretinal fibrosis
* History of Cataract surgey less than 6 months
* History of Glaucoma Surgery ,Vitreoretinal surgery
* Media opacity

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Macular Thickness | 1 month
  Spectral Domain Optical Coherence Tomography

SECONDARY OUTCOMES:
Visual acuity | 1 month
  Early Treatment Diabetic Retinopathy Study

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran